CLINICAL TRIAL: NCT07199452
Title: An Open-Label Clinical Study to Evaluate the Effects of Multiple Oral Doses of Rifabutin on the Single-Dose Pharmacokinetics of MK-4646 in Healthy Participants
Brief Title: A Study of Rifabutin and MK-4646 in Healthy Participants (MK-4646-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 4646-004; MK-4646-004 (Other: MSD)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-4646 (Experimental): On Period 1 Day 1, a single oral dose of MK-4646 will be administered.
  Interventions: Drug: MK-4646
- MK-4646 with Rifabutin (Experimental): Rifabutin will be administered orally once daily from Period 2 Day 1 through Period 2 Day 16. A single oral dose of MK-4646 will be administered on Period 2 Day 14.
  Interventions: Drug: MK-4646; Drug: Rifabutin

INTERVENTIONS:
Drug: MK-4646 — Oral Capsule
Drug: Rifabutin — Oral Capsule
  Arms: MK-4646 with Rifabutin

SUMMARY:
Researchers have designed a new study medicine called MK-4646 as a new way to treat human immunodeficiency virus (HIV). Rifabutin is a medication used to treat tuberculosis (TB).

Researchers want to learn about MK-4646 when taken at the same time as Rifabutin.

They want to:

Measure a person's blood to find out if the amount of MK-4646 in the blood is the same when MK-4646 is taken alone or with Rifabutin Learn about the safety of MK-4646 when taken alone or with Rifabutin and if people tolerate it

ELIGIBILITY:
The main inclusion criteria include but are not limited to:

* Is in good health
* Has a body-mass index (BMI) between 18 and 32 kg/m2

The main exclusion criteria include but are not limited to:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-10-28 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of MK-4646 in Plasma | At designated timepoints (up to approximately 3 days post dose)
  Blood samples will be collected to determine the AUC0-inf of MK-4646 in plasma.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 5 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (1):
- Fortea CRU Madison ( Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com